CLINICAL TRIAL: NCT03067194
Title: Open-label, Multicenter, Randomized Study to Assess the Efficacy and Safety of Celecoxib 200mg Capsule QD and Celecoxib 100mg BID in Hand Osteoarthritis Patients
Brief Title: The Study to Evaluate Efficacy and Safety of Celecoxib Capsule in Hand Osteoarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 266HOA16008
Record Dates: First submitted 2017-02-03; First posted 2017-03-01 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis Hand
Keywords: Osteoarthritis Hand
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib 100mg (Active Comparator): Celecoxib 100mg, Oral, BID(twice per day), During 6 weeks
  Interventions: Drug: Celecoxib 100 MG
- Celecoxib 200mg (Active Comparator): Celecoxib 200mg, Oral, QD(once daily), During 6 weeks
  Interventions: Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: Celecoxib 100 MG — Celecoxib 100mg, Oral, BID(twice per day), During 6 weeks
  Other Names: Celecoxib 100mg capsule
  Arms: Celecoxib 100mg
Drug: Celecoxib 200mg — Celecoxib 200mg, Oral, QD(once daily), During 6 weeks
  Other Names: Celecoxib 200mg capsule
  Arms: Celecoxib 200mg

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Celecoxib capsule in hand osteoarthritis patients.

DETAILED DESCRIPTION:
This is a six-weeks, open-label, multi-center, randomized study. Patients take Celecoxib 200mg capsule once a day or Celecoxib 100mg capsules twice per day. If patients do not tolerate the pain, they are able to take Acetaminophen as a rescue medication during 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Agreement with written informed consent and 19 years of age and older
* Patients history of OA of hand according to ACR criteria
* The 100mm Pain VAS is over 40mm

Exclusion Criteria:

* History of OA of hand surgery
* Intra-articular injections within 3 months
* History of OA of hand infections within 3 months
* Who had taken a drug that has a control of result in clinical trial by investigator's decision
* Pregnant women, nursing mothers or Fertile women who not practice contraception with appropriate methods
* clinically significant hepatic, renal, cardiovascular diseases
* Any history of adverse reaction to the study drugs
* Patients with gastrointestinal ulcers or bleeding disorders
* Finger joint injury within 6 months
* Who had following results after examination

  1. K ≥ 5.5mEq/L
  2. eGFR ≤ 30ml/min/1.73m^2
* Patients on any other clinical trial or experimental treatment in the past 3 months
* Taking narcotic analgesics or patches
* History of drug abuse or alcoholism
* Who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders
* An impossible one who participates in clinical trial by investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
The change of 100mm Pain VAS score at 6 weeks relative to the baseline value of each group | baseline, 6weeks

SECONDARY OUTCOMES:
Changes in each item of K-AUSCAN at 6 weeks relative to the baseline value of each group | baseline, 6weeks
The total point change of K-AUSCAN at 6 weeks relative to the baseline value of each group | baseline, 6weeks
Total score change of insomnia severity at 6 weeks relative to the baseline value of each group | baseline, 6weeks
Total dosing days of acetaminophen for 6 weeks in each group | 6weeks
The total dose of acetaminophen for 6 weeks in each group | 6weeks
Percentage of subjects using acetaminophen for 6 weeks in each group | 6weeks

OTHER OUTCOMES:
Safety assessed by the incidence of adverse event | up to 6weeks
laboratory test(Hematology test, Blood chemistry test, Urinalysis) | up to 6weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Sook Kim, Principal Investigator — Soonchunhyang University Hospital; Chan Hong Jeon, Principal Investigator — Soonchunhyang University Hospital; Sung Hae Jang, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soon Chun Hyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided